CLINICAL TRIAL: NCT04157517
Title: An Open-Label, Dose-Escalation Phase 1b/2 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of Modakafusp Alfa (TAK-573) as a Single Agent and in Combination With Pembrolizumab in Adult Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study of Modakafusp Alfa (TAK-573) Given by Itself and Together With Pembrolizumab in Adults With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to futility.
Sponsor: Teva Branded Pharmaceutical Products R&D LLC (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-573-1001; U1111-1238-9163 (Registry Identifier: WHO)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms; Melanoma
Keywords: Drug Therapy
MeSH Terms: conditions — Neoplasms; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1b SA Dose Escalation (Experimental): Modakafusp alfa 0.1 to 6 milligram per kilogram (mg/kg), infusion, intravenously, once on Day 1 of each 21-days treatment cycle for up to 1 year.
  Interventions: Drug: Modakafusp Alfa
- Phase 2 Safety Lead-in Dose Expansion: Modakafusp Alfa + Pembrolizumab (Experimental): Melanoma with primary resistance to prior anti-PD1, acquired resistance to prior anti-PD1 or naïve to anti-PD1.
  Modakafusp alfa, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once every 6 weeks for up to 2 years. The starting dose of modakafusp alfa for dose expansion safety lead-in phase will be the RP2D determined in the previous Phase 1b dose escalation phase.
  Interventions: Drug: Modakafusp Alfa; Drug: Pembrolizumab
- Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma With Primary Resistance) (Experimental): Melanoma With Primary Resistance to prior anti-PD1. Modakafusp alfa, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once every 6 weeks for up to 2 years, in participants with unresectable/metastatic cutaneous melanoma with primary resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting. The dose of modakafusp alfa for dose expansion phase will be the modakafusp alfa RP2D in combination with pembrolizumab determined in the previous Phase 2 dose expansion safety-lead in phase.
  Interventions: Drug: Modakafusp Alfa; Drug: Pembrolizumab
- Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma With Acquired Resistance) (Experimental): Melanoma With Acquired Resistance to prior anti-PD1. Modakafusp alfa, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once every 6 weeks for up to 2 years, in participants with unresectable/metastatic cutaneous melanoma with acquired resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting. The dose of modakafusp alfa for dose expansion phase will be the modakafusp alfa RP2D in combination with pembrolizumab determined in the previous Phase 2 dose expansion safety lead-in phase.
  Interventions: Drug: Modakafusp Alfa; Drug: Pembrolizumab
- Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma naïve to anti-PD1) (Experimental): Modakafusp alfa, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once every 6 weeks for up to 2 years, in participants with unresectable/metastatic cutaneous melanoma naive to prior line of anti-PD1 containing treatments in the metastatic setting. The dose of modakafusp alfa for dose expansion phase will be the modakafusp alfa RP2D in combination with pembrolizumab determined in the previous Phase 2 dose expansion safety lead-in phase.
  Interventions: Drug: Modakafusp Alfa; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Modakafusp Alfa — Modakafusp alfa intravenous infusion.
  Other Names: TAK-573
Drug: Pembrolizumab — Pembrolizumab intravenous infusion.
  Arms: Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma With Acquired Resistance); Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma With Primary Resistance); Phase 2 Dose Expansion: Modakafusp Alfa + Pembrolizumab (Melanoma naïve to anti-PD1); Phase 2 Safety Lead-in Dose Expansion: Modakafusp Alfa + Pembrolizumab

SUMMARY:
This study has 2 phases.

The main aims of Phase 1b are:

* to check for side effects from modakafusp alfa in adults with locally advanced or metastatic solid tumors.
* to learn how much modakafusp alfa adults can receive without getting any major side effects from it.

The main aims of Phase 2 are:

* to check for side effects from modakafusp alfa when given together with pembrolizumab in adults with metastatic cutaneous melanoma which cannot be completely removed by surgery.
* to learn how these medicines improve their symptoms.

Participants will receive modakafusp alfa for up to 1 year (Phase 1b) or modakafusp alfa given together with pembrolizumab for up to 2 years (Phase 2). Those whose symptoms improve might continue treatment for longer.

In both phases of the study, participants will revisit the study clinic within 30 days after their last dose or before they start other cancer treatment, whichever happens first.

DETAILED DESCRIPTION:
The drug being tested in this study is called modakafusp alfa (TAK-573). Modakafusp alfa is being tested to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and antitumor activity as single agent (SA) or in combination with pembrolizumab in participants with locally advanced or metastatic solid tumors. The study will consist of 2 phases: Phase 1b dose escalation and a Phase 2 dose expansion.

The study will enroll approximately 114 participants (approximately 30 participants in Phase 1b dose escalation phase; 3-9 participants in safety-lead in and 25 participants for each expansion cohort (3 cohorts) of Phase 2.

The dose escalation phase will enroll participants with solid tumors. The dose escalation phase is to evaluate SA recommended phase 2 dose (RP2D).

The dose expansion phase in combination with pembrolizumab will be initiated with a safety lead-in phase once the SA RP2D is determined for modakafusp alfa. The dose expansion will include participants with one of following 3 disease indications:

I. Unresectable/metastatic cutaneous melanoma with primary resistance to no more than 2 prior lines of anti-disease programmed cell death protein 1 (PD1) containing treatments in the metastatic setting.

II. Unresectable/metastatic cutaneous melanoma with acquired resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting.

III. Unresectable/metastatic cutaneous melanoma naïve to prior anti-PD1 containing treatments in the metastatic setting.

This multi-center trial will be conducted in the United States and Australia. Participants with demonstrated clinical benefit may continue treatment beyond 1 year for Phase 1b and 2 years for Phase 2 if approved by the sponsor. The overall time to participate in this study is 55 months. All participants will make an end of treatment (EOT) visit 30 days after receiving their last dose of study drug or before the start of subsequent systemic anticancer therapy, whichever occurs first for a safety follow up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
2. For both the dose escalation and expansion cohort phases of the study, eligible participants must have histologically confirmed advanced (locoregionally recurrent, not amenable to curative therapy) or metastatic solid tumors.
3. Measurable disease per RECIST v1.1. At least 1 target lesion amenable for biopsy is required for enrollment in phase 1b. A minimum of 1 target lesion for response assessment is required for enrollment in phase 2. A separate lesion amenable for biopsy is required for enrollment in phase 2 for cohorts I and II post futility analysis and for all participants (safety lead-in and expansion) with subgroup III melanoma.
4. Phase 1b Dose Escalation: Participants with histologically confirmed advanced locally (locoregionally recurrent, not amenable to curative therapy) or metastatic solid tumors.

Phase 2 Dose Expansion:

The combination cohorts, including participants in the safety-lead phase, will enroll participants with unresectable/metastatic melanoma in the following subgroups:

I. Unresectable/metastatic histologically confirmed cutaneous melanoma with primary resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting.

II. Unresectable/metastatic histologically confirmed cutaneous melanoma with acquired resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting.

III. Unresectable/metastatic histologically confirmed cutaneous melanoma naive to prior anti-PD1 containing treatments in the metastatic setting.

* Participants with BRAF V600E mutant melanoma may have received prior BRAF inhibitor therapy.
* For the expansion cohorts I and II, there is no limitation of total number of prior line(s) of therapy, but the number of prior line(s) containing anti-PD1 must be ≤2 in the metastatic setting.
* For the expansion cohort III, participants who received an anti-PD-1 treatment in the adjuvant setting must have completed that treatment at least 6 months prior to enrollment and must not have progressed on the anti-PD1 adjuvant treatment.
* Primary resistance is defined as a best response of PD or SD less than (<) 6 months to an anti-PD1 alone or in combination with other agents (that is, CTLA4) in the initial anti-PD1 containing treatment.
* Acquired resistance is defined as a progression following a best response of CR, PR or SD>6 months to a prior anti-PD1 alone or in combination with other agents (that is, CTLA4).

Exclusion Criteria:

1. Persistent toxicity from previous treatments that has not resolved to less than or equal to (<=) CTCAE version 5.0 Grade 1 prior to administration of modakafusp alfa, except for alopecia, Grade 2 neuropathy, and Grade 2 asthenia/fatigue, or autoimmune endocrinopathies with stable replacement therapy.
2. History of any of the following <=6 months before first dose modakafusp alfa: New York Heart Association (NYHA) Grade III or IV congestive heart failure, unstable angina, myocardial infarction, unstable symptomatic ischemic heart disease, any ongoing symptomatic cardiac arrhythmias of Grade >2, pulmonary embolism, or symptomatic cerebrovascular events, or any other serious cardiac condition (example, symptomatic pericardial effusion or restrictive cardiomyopathy). Chronic, stable atrial fibrillation on stable anticoagulant therapy, including low molecular-weight heparin, is allowed.
3. Baseline QT interval with Fridericia's correction (QTcF) greater than (>) 480 millisecond (msec) (Grade >=2), history of congenital long QT syndrome, or torsades de pointes.
4. Patients with acral lentiginous melanoma are excluded in phase 2 except for the safety lead-in phase.
5. Ongoing or active infection.
6. Known history of human immunodeficiency virus (HIV) infection or any other relevant congenital or acquired immunodeficiency. Testing during screening period is required only if indicated by specific local regulations or investigator's criteria.
7. Known hepatitis B (HBV) surface antigen seropositive or detectable hepatitis C infection viral load. Note: Participants with a positive HBV core antibody can be enrolled but must have an undetectable hepatitis B viral load.
8. Autoimmune disease requiring systemic immunosuppressive therapy. Participants with immune mediated endocrine deficiency from previous therapy with stable hormone replacement are exceptions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (15):
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - The Angeles Clinic and Research Institute - West Los Angeles Office, Los Angeles, California
  - University of Colorado Health Memorial Hospital Central, Colorado Springs, Colorado
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Norris Cotton Cancer Center Lebanon, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Intermountain Medical Center, Murray, Utah
  - West Virginia University Health Sciences Campus, Morgantown, West Virginia
- Australia (2):
  - The Queen Elizabeth Hospital, Woodville South, South Australia
  - Ballarat Regional Integrated Cancer Center, Ballarat, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be assessed for scientific merit, product approval status, and conflicts of interest. If the request is approved, patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please visit USMedInfo@tevapharm.com to make your request.

REFERENCES:
- [Derived] Gill D, Cowey CL, Daniels GA, Sommerhalder D, Abdul-Karim R, Kirkwood JM, Kolodney J, Mehmi I, Roberts-Thomson R, Strauss J, Thomas S, Whitman E, Xing Y, McKean M, Collins S, Li C, Saggu G, Chen T, Wang S, Lewis M, Parot X, Johnson M. A phase Ib/II study of modakafusp alfa alone and in combination with pembrolizumab in patients with advanced or metastatic solid tumors. Front Oncol. 2025 Dec 8;15:1620987. doi: 10.3389/fonc.2025.1620987. eCollection 2025. PMID 41445795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 17 investigative sites in the United States and Australia from 12 December 2019 to 20 December 2023.
Pre-assignment Details: Participants were enrolled to Phase 1b (Dose Escalation) to receive single agent modakafusp alfa, and combination therapy of modakafusp alfa and pembrolizumab in Phase 2 (Safety lead-in, and Expansion with 3 Cohorts [Cohorts I, II and III). Cohort III had no enrolment due to strategic reason, therefore, no data was collected and reported for Cohort III in this report.
Groups:
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 0.1 milligrams per kilogram (mg/kg), infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 0.2 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 0.4 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 0.75 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 1.5 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg: Participants with any of the 3-melanoma disease of expansion Cohort I, II or III received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
- Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg: Participants with unresectable/metastatic cutaneous melanoma with primary resistance to no more than 2 prior lines of anti- programmed cell death protein 1 (PD1) containing treatments in the metastatic setting received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
- Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg: Participants with unresectable/metastatic cutaneous melanoma with acquired resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
- Phase 2, Expansion, Cohort III: Modakafusp Alfa + Pembrolizumab: Participants with unresectable/metastatic cutaneous melanoma naïve to prior line of anti-PD1 containing treatments in the metastatic setting were planned to receive modakafusp alfa, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
Period: Overall Study
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort III: Modakafusp Alfa + Pembrolizumab
Started | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 9 | 12 | 0 (No participants were enrolled in Cohort III due to strategic reason.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 9 | 12 | 0
Not completed — Death | 1 | 2 | 2 | 3 | 3 | 4 | 1 | 2 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 7 | 7 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all enrolled participants who received at least one dose (even incomplete) of modakafusp alfa.
Groups:
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg: Participants with advanced/metastatic tumors received modakafusp alfa 0.1 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Total: Total of all reporting groups
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 9 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.0 (5.20) | 51.3 (11.37) | 68.0 (10.44) | 62.0 (8.19) | 55.0 (4.58) | 61.8 (9.13) | 74.3 (4.04) | 53.4 (17.91) | 60.3 (12.11) | 60.7 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 1 | 2 | 4 | 2 | 4 | 1 | 16
  Male | 2 | 2 | 3 | 2 | 1 | 2 | 1 | 5 | 11 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 7
  Not Hispanic or Latino | 3 | 2 | 2 | 2 | 1 | 5 | 2 | 8 | 8 | 33
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 3 | 2 | 3 | 2 | 5 | 3 | 8 | 9 | 38
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b and Phase 2 Safety Lead-in: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: Adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment. A TEAE was any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: From signing of the informed consent form (ICF) through 30 days after last dose of study drug or the start of subsequent anticancer therapy, whichever occurred first (up to 1 year 1 month for Phase 1b and 2 years 1 month for Phase 2)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants | 3 | 3 | 3 | 3 | 3 | 6 | 3

2. Primary Outcome: Phase 1b and Phase 2 Safety Lead-in: Number of Participants With Grade 3 or Higher TEAEs
Description: TEAEs Grades were evaluated as per the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0. (NCI CTCAE v5), where Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living (ADL). Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE.
Time Frame: From signing of the ICF through 30 days after last dose of study drug or the start of subsequent anticancer therapy, whichever occurred first (up to 1 year 1 month for Phase 1b and 2 years 1 month for Phase 2)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants | 2 | 1 | 2 | 2 | 3 | 4 | 2

3. Primary Outcome: Phase 1b and Phase 2 Safety Lead-in: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following AEs that occurred in the escalation phase or in the combination safety lead-in phase during Cycle 1 unless they were considered by the investigator to be clearly unrelated to therapy with modakafusp alfa according to NCI CTCAE version 5.0. Any Grade 5 TEAE. Febrile neutropenia: Grade >=3 or 4 neutropenia. Grade 4 thrombocytopenia. Grade >=3 thrombocytopenia. Any Grade 3 immune-related AEs such as pericarditis, pneumonitis, cardiotoxicity, hepatitis, or neurotoxicity. Delay in the initiation of Cycle 2 by more than 14 days from the calculated start date due to a lack of adequate recovery of treatment-related hematological or nonhematologic toxicities. Any Grade >=3 nonhematologic toxicity with some exception. Any Grade 2 nonhematologic toxicity that was considered by the investigator to be related to study drug and dose-limiting.
Time Frame: Cycle 1 (Cycle length is equal to [=] 21 days)
Population: DLT evaluable analysis set included participants who received all Cycle 1 doses of modakafusp alfa or experience a DLT in Cycle 1 in the dose-escalation portion of the study; or participants who received all Cycle 1 doses of modakafusp alfa in combination with pembrolizumab or experience a DLT in Cycle 1 in the safety lead-in portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 0

4. Primary Outcome: Phase 1b and Phase 2 Safety Lead-in: Number of Participants Reporting One or More Serious Adverse Event (SAEs)
Description: SAE was defined as any untoward medical occurrence that resulted in death; was life-threatening; required inpatient hospitalization or prolongation of an existing hospitalization; resulted in persistent or significant disability or incapacity; was a congenital anomaly/birth defect; was a medically important event that might not result in death, be immediately life-threatening, or required hospitalization, but might be considered serious when, on the basis of appropriate medical judgment, it might jeopardize the participant, required medical or surgical intervention to prevent one of the outcomes listed above, or involves suspected transmission via a medicinal product of an infectious agent.
Time Frame: From signing of the ICF through 30 days after last dose of study drug even if the participants start non-protocol systemic therapy (up to 1 year 1 month for Phase 1b and 2 years 1 month for Phase 2)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants | 3 | 1 | 2 | 1 | 2 | 4 | 0

5. Primary Outcome: Phase 1b and Phase 2 Safety Lead-in: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuations
Description: TEAE was defined as any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: as for outcome 2
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
Participants
  TEAEs Leading to Dose Modifications | 0 | 0 | 2 | 1 | 1 | 4 | 1
  TEAEs Leading to Treatment Discontinuations | 0 | 0 | 1 | 0 | 0 | 2 | 0

6. Primary Outcome: Phase 2 Expansion: Overall Response Rate (ORR) Based on RECIST v1.1
Description: ORR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR: At least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose of study drug up to end of treatment or end of study (up to 2 years)
Population: The response evaluable analysis set included participants with measurable disease at baseline and at least 1 post-treatment evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
percentage of participants | 0.0 [0.0 to 33.6] | 16.7 [2.1 to 48.4]

7. Secondary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) of Modakafusp Alfa
Description: The MTD was selected as the highest dose which has maximum probability of being in targeted toxicity interval.
Time Frame: Cycle 1 (Cycle length = 21 days)
Population: DLT evaluable analysis set included participants who received all Cycle 1 doses of modakafusp alfa or experience a DLT in Cycle 1 in the dose-escalation portion of the study.
Measure: Number; unit: milligrams per kilograms (mg/kg)
Groups:
- Phase 1b, Dose Escalation: All Participants: All participants with advanced/metastatic tumors in Phase 1b who received modakafusp alfa 0.1, 0.2, 0.75, 1.0 or 1.5 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
Arm/Group | Phase 1b, Dose Escalation: All Participants
Number analyzed (Participants) | 21
milligrams per kilograms (mg/kg) | NA — MTD was not determined because criteria was not met.

8. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Recommended Phase 2 Dose (RP2D) for Single Agent (SA) Modakafusp Alfa in Phase 1b and in Combination With Pembrolizumab in Phase 2 Safety Lead-in
Description: The RP2D of modakafusp alfa as a single agent or in combination with pembrolizumab was determined based on safety (including DLTs), pharmacokinetic and clinical data. DLT was graded according to CTCAE v5.0.
Time Frame: Cycle 1 (Cycle length = 21 days)
Population: as for baseline characteristics
Measure: Number; unit: mg/kg
Arm/Group | Phase 1b, Dose Escalation: All Participants | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 21 | 3
mg/kg | 1.0 | 1.0

9. Secondary Outcome: Phase 2 Expansion: Number of Participants Reporting One or More TEAEs
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence did not necessarily have a causal relationship with this treatment. A TEAE was any AE either reported for the first time or worsening of a pre-existing event after first dose of study drug and within 30 days of the last administration of study drug.
Time Frame: From signing of the ICF through 30 days after last dose of study drug or the start of subsequent anticancer therapy, whichever occurred first (up to 2 years 1 month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
Participants | 8 | 12

10. Secondary Outcome: Phase 2 Expansion: Number of Participants With Grade 3 or Higher TEAEs
Description: as for outcome 2
Time Frame: as for outcome 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
Participants | 6 | 7

11. Secondary Outcome: Phase 2 Expansion: Number of Participants Reporting One or More SAEs
Description: as for outcome 4
Time Frame: From signing of the ICF through 30 days after last dose of study drug even if the participants start non-protocol systemic therapy (up to 2 years 1 month)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
Participants | 2 | 6

12. Secondary Outcome: Phase 2 Expansion: Number of Participants With One or More TEAEs Leading to Dose Modifications and Treatment Discontinuations
Description: as for outcome 5
Time Frame: as for outcome 9
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
Participants
  TEAEs Leading to Dose Modifications | 1 | 9
  TEAEs Leading to Treatment Discontinuations | 0 | 1

13. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Maximum Observed Serum Concentration (Cmax) for Modakafusp Alfa
Description: Cmax for modakafusp alfa was reported.
Time Frame: Phase 1b, Cycles 1 and 2 Day 1: Pre-infusion and at multiple timepoints (up to 72 hours) post-infusion; Phase 2, Safety lead-in, Cycles 1 and 3 Day 1: Pre-infusion and at multiple timepoints (up to 72 hours) post-infusion (each cycle length=21 days)
Population: Pharmacokinetic (PK) analysis set included participants who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. As planned, PK data at Cycles 1 and 2 Day 1 for Phase 1b, and Cycles 1 and 3 Day 1 for Phase 2 (Safety lead-in) was reported. Here, "number analyzed" signified participants who were evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
nanograms per milliliter (ng/mL)
  Cycle 1 Day 1 | 261 (85.0) | 2770 (51.4) | 4920 (42.9) | 17000 (26.1) | 17700 (60.1) | 37200 (29.9) | 21200 (18.7)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2 | 3 | 0
  Cycle 2 Day 1 | 336 (540.2) | 2790 (14.2) | 3560 (99.9) | 9420 (52.7) | 14400 (136.2) | 25400 (84.5) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 13900 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

14. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Time to Reach the Cmax (Tmax) for Modakafusp Alfa
Description: Tmax for modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: PK analysis set included participants who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. As planned, PK data at Cycles 1 and 2 Day 1 for Phase 1b, and Cycles 1 and 3 Day 1 for Phase 2 (Safety lead-in) was reported. Here, "overall number of participants analyzed" signified participants who were evaluable for this outcome measure and "number analyzed" signified participants who were evaluable at specified timepoints.
Measure: Median (Full Range); unit: hour
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3
hour
  Cycle 1 Day 1 | 1.53 [1.48 to 1.72] | 1.17 [1.03 to 1.17] | 1.05 [0.98 to 1.20] | 1.18 [1.17 to 2.12] | 1.52 [1.12 to 2.02] | 1.97 [1.03 to 2.72] | 3.13 [2.60 to 3.42]
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2 | 3 | 0
  Cycle 2 Day 1 | 1.28 [1.05 to 1.50] | 1.03 [1.00 to 1.05] | 1.05 [0.92 to 3.92] | 1.07 [1.03 to 3.18] | 1.77 [1.60 to 1.93] | 1.97 [1.03 to 2.72] |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 2.90 [2.90 to 2.90]

15. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Area Under the Plasma Concentration-time Curve From Time 0 to Last Measurable Concentration (AUClast) for Modakafusp Alfa
Description: AUClast for modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: PK analysis set included participants who had sufficient data to calculate at least 1 PK parameter for modakafusp alfa. As planned, PK data at Cycles 1 and 2 Day 1 for Phase 1b, and Cycles 1 and 3 Day 1 for Phase 2 (Safety lead-in) was reported. Here, "number analyzed" signified participants who were evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 3 | 2 | 3 | 6 | 3
  Cycle 1 Day 1 | 458 (135.8) | 8450 (70.0) | 33100 (72.4) | 183000 (74.1) | 262000 (61.5) | 897000 (57.1) | 455000 (21.8)
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 2 | 3 | 3 | 2 | 2 | 0
  Cycle 2 Day 1 | 535 (1101.2) | 8030 (9.3) | 20300 (153.2) | 86300 (81.7) | 159000 (219.2) | 360000 (112.5) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 165000 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

16. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) for Modakafusp Alfa
Description: AUCinf of modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 6 | 3
h*ng/mL
  Cycle 1 Day 1 | 1470 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 8780 (66.3) | 33100 (72.2) | 217000 (60.2) | 263000 (61.5) | 1060000 (62.1) | 455000 (21.8)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 3 | 3 | 2 | 0
  Cycle 2 Day 1 | 2540 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 8840 (7.1) | 21100 (140.1) | 86400 (81.6) | 160000 (218.7) | 372000 (121.3) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 165000 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

17. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Terminal Disposition Phase Half-life (t1/2z) for Modakafusp Alfa
Description: T1/2z of modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 6 | 3
hour
  Cycle 1 Day 1 | 1.07 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 1.97 (33.9) | 5.25 (13.7) | 5.60 (28.5) | 6.23 (14.4) | 15.5 (71.8) | 6.44 (11.0)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 3 | 0
  Cycle 2 Day 1 | 0.832 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 1.85 (9.1) | 3.08 (38.6) | 6.43 (11.3) | 6.15 (7.7) | 14.1 (85.6) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 6.15 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

18. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Total Clearance (CL) After Intravenous Administration for Modakafusp Alfa
Description: CL was total clearance of the drug from the serum. CL of modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour per kilograms (L/h/kg)
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 6 | 3
liters per hour per kilograms (L/h/kg)
  Cycle 1 Day 1 | 0.0682 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 0.0228 (66.2) | 0.0121 (72.4) | 0.00345 (61.0) | 0.00383 (61.1) | 0.00142 (61.1) | 0.00220 (21.3)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 2 | 0
  Cycle 2 Day 1 | 0.0394 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 0.0226 (7.2) | 0.0190 (139.6) | 0.00872 (81.1) | 0.00632 (214.5) | 0.00407 (118.5) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 0.00610 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

19. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: Volume of Distribution at Steady State (Vss) for Modakafusp Alfa
Description: Vss of modakafusp alfa was reported.
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per kilograms (L/kg)
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg
Number analyzed (Participants) | 1 | 3 | 3 | 3 | 3 | 6 | 3
liters per kilograms (L/kg)
  Cycle 1 Day 1 | 0.119 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 0.0567 (49.7) | 0.0562 (58.2) | 0.0276 (13.5) | 0.0369 (48.1) | 0.0331 (33.1) | 0.0313 (13.3)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 3 | 2 | 2 | 0
  Cycle 2 Day 1 | 0.0546 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant. | 0.0565 (15.6) | 0.0794 (135.8) | 0.0562 (72.9) | 0.0514 (107.2) | 0.0629 (33.4) |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  | 0.0453 (NA) — Here "NA" means Geometric Coefficient of Variation could not be calculated for a single participant.

20. Secondary Outcome: Phase 1b and Phase 2 Safety Lead-in: ORR Based on RECIST v1.1
Description: ORR was defined as the percentage of participants who achieved CR or PR as per RECIST version 1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose of study drug up to end of treatment or end of study (up to 1 year for Phase 1b and 2 years for Phase 2)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400mg: Participants with any of the 3-melanoma disease of expansion Cohort I, II or III received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400mg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 4 | 3
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]

21. Secondary Outcome: Phase 1b and Phase 2: Disease Control Rate (DCR) Based on RECIST v1.1
Description: DCR was defined as the percentage of participants who achieved CR, PR, or stable disease (SD) (determined by the investigator) as per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression (PD), taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 20
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 2 | 4 | 3 | 9 | 12
percentage of participants | 0 [0.0 to 84.2] | 50.0 [1.3 to 98.7] | 0 [0.0 to 84.2] | 33.3 [0.8 to 90.6] | 0 [0.0 to 84.2] | 50.0 [6.8 to 93.2] | 33.3 [0.8 to 90.6] | 33.3 [7.5 to 70.1] | 41.7 [15.2 to 72.3]

22. Secondary Outcome: Phase 1b and Phase 2: Duration of Response (DOR) Based on RECIST v1.1
Description: DOR was defined as the time from the first documentation of a response (CR or PR) until PD or death, whichever occurred first as per RECIST v1.1. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From the date of first documentation of a CR or PR until PD or death, whichever occurred first (up to end of treatment or end of study [1 year for Phase 1b and 2 years for Phase 2])
Population: The response evaluable analysis set included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Here, "overall number of participants analyzed" signified participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
months |  |  |  |  |  |  |  |  | NA [NA to NA] — Here "NA" means median and 95% confidence interval could not be estimated due to insufficient events.

23. Secondary Outcome: Phase 1b and Phase 2: Time to Progression (TTP) Based on RECIST v1.1
Description: TTP was defined as the time from the date of the first dose of study drug to the date of the first documentation of PD according to RECIST v1.1. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From the date of the first dose of study drug to the date of the first documentation of PD (up to end of treatment or end of study [1 year for Phase 1b and 2 years for Phase 2])
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 1 | 4 | 3 | 8 | 7
months | 2.4 [1.41 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 4.5 [1.41 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.7 [0.79 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.4 [1.38 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.5 [NA to NA] — Here "NA" means upper and lower limits of 95% confidence interval could not be estimated due to insufficient events. | 2.3 [1.35 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.7 [1.31 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 2.8 [1.28 to 6.01] | 2.3 [1.35 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events.

24. Secondary Outcome: Phase 1b and Phase 2: Progression Free Survival (PFS) Based on RECIST v1.1
Description: PFS was defined as the time from the date of the first dose of study drug to the date of first documentation of PD according to RECIST v.1.1, or death due to any cause, whichever occurred first. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: From the date of the first dose of study drug to the date of first documentation of PD or death, whichever occurred first (up to end of treatment or end of study [1 year for Phase 1b and 2 years for Phase 2])
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 9 | 12
months | 2.4 [1.41 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.6 [1.41 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.7 [0.79 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.4 [1.38 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.8 [1.48 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.9 [0.95 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 1.7 [1.31 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 4.8 [1.31 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 2.6 [1.38 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events.

25. Secondary Outcome: Phase 1b and Phase 2: Overall Survival (OS) Based on RECIST v1.1
Description: OS was defined as the time from the date of first dose of study drug to the date of death due to any cause.
Time Frame: From the date of first dose of study drug to the date of death due to any cause (up to end of treatment or end of study [1 year for Phase 1b and 2 years for Phase 2])
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 3 | 9 | 12
months | NA [3.61 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events. | 9.8 [1.64 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 7.0 [0.99 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 6.3 [2.99 to NA] — Here "NA" means the upper limit of 95% confidence interval could not be estimated due to small number of death events resulting large variability and therefore the upper 95% confidence limits of Kaplan-Meier survival estimate remaining above 50%. | 4.3 [1.84 to NA] — Here "NA" means the upper limit of 95% confidence interval could not be estimated due to small number of death events resulting large variability and therefore the upper 95% confidence limits of Kaplan-Meier survival estimate remaining above 50%. | 3.1 [0.95 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | NA [5.13 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events. | NA [5.62 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events. | NA [2.60 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events.

26. Secondary Outcome: Phase 2 Expansion: ORR Based on Based on Immune Response Evaluation Criteria in Solid Tumors (iRECIST)
Description: ORR was defined as the percentage of participants whose BOR was immune CR (iCR) or immune PR (iPR), according to iRECIST as per investigator assessment. iCR: immune complete response achieved with disappearance of all target lesions immune confirmed progressive disease (iCPD). (iCPD): immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. iSD: immune stable disease in the absence of iCR or immune PD (iPD). iUPD: immune unconfirmed progressive disease (iUPD) when iCPD is unconfirmed NE: not evaluable.
Time Frame: From date of first dose of study drug until confirmed iCR or iPR (up to end of treatment or end of study [up to 2 years])
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 8 | 12
percentage of participants | 0.0 [0.0 to 36.9] | 16.7 [2.1 to 48.4]

27. Secondary Outcome: Phase 2 Expansion: DCR Based on iRECIST
Description: DCR was defined as percentage of participants who have achieved the best response of iCR, iPR, iSD based on iRECIST as per investigator assessment. iCR: achieved with disappearance of all target lesions, iPR: achieved with disappearance of partial target lesions. iSD: in the absence of iCR or iCPD. iUPD: when iPD is unconfirmed NE: not evaluable.
Time Frame: as for outcome 26
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg: Participants with unresectable/metastatic cutaneous melanoma with primary resistance to no more than 2 prior lines of PD1 containing treatments in the metastatic setting received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 8 | 12
percentage of participants | 37.5 [8.5 to 75.5] | 41.7 [15.2 to 72.3]

28. Secondary Outcome: Phase 2 Expansion: DOR Based on iRECIST
Description: DOR was defined as time from date of first observation of response (iPR or iCR) to date of the first observation of progression (iCPD) based on iRECIST as per investigator assessment, or date of death, whatever the cause. iCR: immune complete response achieved with disappearance of all target lesions iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first documented confirmed iCR or iPR until first documentation of iCPD or death (up to end of treatment or end of study [up to 2 years])
Population: The response evaluable analysis set included participants with measurable disease at baseline and at least 1 post-treatment evaluation. Here, "overall number of participants analyzed" signifies participants who had iCR or iPR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 0 | 2
months |  | NA [NA to NA] — Here "NA" means median and 95% confidence interval could not be estimated due to insufficient events.

29. Secondary Outcome: Phase 2 Expansion: TTP Based on iRECIST
Description: TTP was defined as the time from the date of the first dose of study drug to the date of the first documentation of iCPD based on iRECIST as per investigator assessment. iCPD: immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From the date of the first dose of study drug to the date of the first documentation of iCPD (up to end of treatment or end of study [up to 2 years])
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
months | 4.8 [1.31 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | NA [1.38 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to insufficient events.

30. Secondary Outcome: Phase 2 Expansion: PFS Based on iRECIST
Description: PFS was defined as the time from the first dose date to the date of iCPD or date of death (whichever occurred first) based on iRECIST as per investigator assessment. iCPD was defined as immune confirmed progressive disease when there is either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dose of study drug until confirmed iCPD or death (up to end of treatment or end of study [up to 2 years])
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 9 | 12
months | 4.8 [1.31 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events. | 2.6 [2.6 to NA] — Here "NA" means upper limit of 95% confidence interval could not be estimated due to insufficient events.

31. Secondary Outcome: Phase 1b and Phase 2: Number of Participants With Positive Anti-Modakafusp Alfa Antibodies (ADA) Status
Description: ADA samples scoring equal to or above the cut-point (titer of 75) were defined as ADA positive.
Time Frame: Baseline up to end of treatment or end of study (up to 1 year for Phase 1b and 2 years for Phase 2)
Population: Immunogenicity-evaluable analysis set included participants with a baseline and at least one post-baseline immunogenicity assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 3 | 9 | 10
Participants | 2 | 2 | 3 | 3 | 3 | 4 | 3 | 9 | 10

32. Secondary Outcome: Phase 1b and Phase 2: Titer of Anti-Modakafusp Alfa Antibodies (ADA)
Description: ADA titers were assessed by confirmatory assay.
Time Frame: Baseline up to end of treatment or end of study (up to 1 year for Phase 1b and 2 years for Phase 2)
Population: as for outcome 31
Measure: Median (Full Range); unit: titers
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp 1.0 mg/kg Alfa + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort I: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg | Phase 2, Expansion, Cohort II: Modakafusp Alfa 1.0 mg/kg + Pembrolizumab 400 mg
Number analyzed (Participants) | 2 | 2 | 3 | 3 | 3 | 4 | 3 | 9 | 10
titers | 150.0 [75 to 225] | 164000.0 [2020 to 1480000] | 6070.0 [675 to 492000] | 6070.0 [75 to 164000] | 6070.0 [2020 to 54700] | 109350.0 [2020 to 492000] | 273350.0 [225 to 1480000] | 492000.0 [225 to 4430000] | 164000.0 [225 to 1480000]

ADVERSE EVENTS:
Time Frame: From signing of the ICF through 30 days after last dose of study drug or the start of subsequent anticancer therapy, whichever occured first (up to 1 year 1 month for Phase 1b and 2 years 1 month for Phase 2)
Groups:
- Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg: Participants received modakafusp alfa 0.1mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle.
- Phase 2, Safety Lead-in: Modakafusp Alfa + Pembrolizumab: Participants with any of the 3-melanoma disease of expansion Cohort I, II or III received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
- Phase 2, Expansion, Cohort I: Modakafusp Alfa + Pembrolizumab: Participants with unresectable/metastatic cutaneous melanoma with primary resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
- Phase 2, Expansion, Cohort II: Modakafusp Alfa + Pembrolizumab: Participants with unresectable/metastatic cutaneous melanoma with acquired resistance to no more than 2 prior lines of anti-PD1 containing treatments in the metastatic setting received modakafusp alfa 1.0 mg/kg, infusion, intravenously, once on Day 1 of each 21-days treatment cycle and pembrolizumab 400 mg infusion, intravenously, once, every 6 weeks.
Arm/Group | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg | Phase 2, Safety Lead-in: Modakafusp Alfa + Pembrolizumab | Phase 2, Expansion, Cohort I: Modakafusp Alfa + Pembrolizumab | Phase 2, Expansion, Cohort II: Modakafusp Alfa + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 2/3 | 3/3 | 3/3 | 4/6 | 1/3 | 2/9 | 4/12
Serious Adverse Events (participants affected / at risk) | 3/3 | 1/3 | 2/3 | 1/3 | 2/3 | 4/6 | 0/3 | 2/9 | 6/12
Other Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 3/3 | 3/3 | 3/3 | 6/6 | 3/3 | 8/9 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg (N=6) | Phase 2, Safety Lead-in: Modakafusp Alfa + Pembrolizumab (N=3) | Phase 2, Expansion, Cohort I: Modakafusp Alfa + Pembrolizumab (N=9) | Phase 2, Expansion, Cohort II: Modakafusp Alfa + Pembrolizumab (N=12)
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 2
Intussusception (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.1 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.2 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.4 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 0.75 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 1.0 mg/kg (N=3) | Phase 1b, Dose Escalation: Modakafusp Alfa 1.5 mg/kg (N=6) | Phase 2, Safety Lead-in: Modakafusp Alfa + Pembrolizumab (N=3) | Phase 2, Expansion, Cohort I: Modakafusp Alfa + Pembrolizumab (N=9) | Phase 2, Expansion, Cohort II: Modakafusp Alfa + Pembrolizumab (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 2 | 1
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
Bell's palsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Blood pressure fluctuation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chills (General disorders) | 3 | 0 | 1 | 1 | 2 | 3 | 0 | 3 | 5
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 4
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 3
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 4 | 7
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 4 | 9
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 6
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Intensive care unit delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 4
Libido decreased (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 3 | 1 | 4 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 3 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 1 | 2 | 4
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Study was terminated early due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-07-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04157517/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT04157517/SAP_001.pdf